CLINICAL TRIAL: NCT06609122
Title: Impact of Animal-Assisted Intervention Dogs on the Performance Behaviors of Special Needs
Brief Title: Impact of AAI Dogs on Performance and Behavior of Children with Autism
Acronym: AAI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wilfred Hing-sang WONG, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW19-131; MHIFS (Other Grant/Funding Number: Mental Health Initiatives Funding, Health Bureau, The Government of the Hong Kong Special Administrative Region); HKU/HA HKW IRB (Other: Hong Kong Hospital Authority)
Record Dates: First submitted 2024-09-10; First posted 2024-09-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Animal Assisted Intervention; Animal Assisted Education; Animal Assisted Therapy; Therapy Dog; Animal Assisted Education Dog; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are unaware of which treatment they are receiving, but the researchers know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Students join the standard class at the same time slot
- Intervention Group (Experimental): The teacher will work on the training goals with incorporation of the dog in the activity. For example, in the training of comprehension of commands, participant would be asked to take one item out of a few items, and then to pass to the dog. If correction of articulation errors is indicated (e.g. misarticulated /k/), training items would be picked under consideration of linkage to dogs. Words like '狗' /kɐu2/ and '教' /kau3/ would be used as stimuli during training.
  Interventions: Other: Animal Assisted Intervention

INTERVENTIONS:
Other: Animal Assisted Intervention — Animal-assisted intervention (AAI) is a therapeutic approach that involves animals as part of a treatment plan to improve physical, social, emotional, or cognitive functioning in individuals. Animals such as dogs, cats, horses, and even dolphins are commonly used in AAI due to their ability to provide comfort, companionship, and motivation.
  AAI can take many forms, including animal-assisted therapy (AAT), where a trained therapy animal works with a licensed healthcare professional to achieve specific treatment goals. Animal-assisted activities (AAA) involve interactions with animals in a more casual and recreational setting, such as visits to hospitals or nursing homes to provide companionship and emotional support.
  Arms: Intervention Group

SUMMARY:
Autism Spectrum Disorder (ASD) is a lifelong neurodevelopmental disorder usually diagnosed in early childhood. Children with ASD exhibit social communication and interaction problems, which may cause deficits in social-emotional reciprocity, problems with developing, maintaining, and understanding relationships, and abnormal nonverbal communicative behaviors such as impaired eye contact and body language. Some children with ASD have severe behavioral problems, such as stereotyped or repetitive motor movements, and extreme distress at small changes. ASD is a complex and individualized disorder, which creates challenges in treatment.

Animal-assisted education (AAE) programmes have been introduced for children with special needs in other countries such as the United States and Australia. PAALS (Palmetto Animal Assisted Life Services) in the United States have introduced the Pet a PAALS Dog programme, which assists stressed students at USC (University of South Carolina). Assistance Dogs Australia has provided an Educational Support Dog Echo to Kalinda Support School, for children with a wide range of disabilities. Existing literature indicate the benefit of animal-assisted therapy on physical, behavioral, and cognitive disabilities, especially in social and communication disorders. Formally trained human-dog teams in animal-assisted interventions (AAI) can play a unique role in social and communicative development that schools, and caregivers may not be able to provide. Interacting with animal-assisted intervention dogs can increase children with ASD&amp;amp;#39;s social interaction, communication, and effective connection. Dogs can also provide emotional support in stressful situations such as calming the child down when they have a tantrum. Moreover, animal-assisted therapy has shown to decrease stress levels, anxiety, and restrictive and repetitive behavior patterns. Dogs as pets can also bring significant improvements to caregivers of children with ASD and improve conflict management.

Based on a successful pilot trial in 2019 with 8 children showed that AAI program has a positive effect on the performance of children with ASD, The investigator proposed an observational study that tracks the effectiveness of an animal-assisted intervention programme in a local school for children with ASD and developmental disabilities.

DETAILED DESCRIPTION:
This is an observational study that tracks the effectiveness of an AAI dog program in a local school for children with ASD and developmental disabilities.

1. To evaluate the effectiveness of AAI on speech and language training, and quality of life in children with autism.
2. To identify any problems of AAI carried out based on this protocol.
3. To evaluate the cost of implementing AAI in Hong Kong.

For the pilot study, two to four students with mild to moderate autism which diagnosed by paediatrician will be selected through the following procedure. The pilot study of the animal-assisted intervention programme consists of two 15-min sessions per week, and a total of 8 sessions will be conducted at the chosen intervention centre from April 2019 to May 2019. The main study will be one year from April 2019 to April 2020. The intervention will occur in both individual and group settings. 2 to 4 students will be allocated to each individual session, and others will attend the group sessions. The project team will be made up of many professional including a qualified AAI dog, qualified AAI dog handler, occupational therapist, pediatrician, clinical psychologist, speech therapist, school teacher or school social worker. For the pilot study, two to four students with mild to moderate autism which diagnosed by paediatrician will be selected through the following procedure. The pilot study of the animal-assisted intervention programme consists of two 15-min sessions per week, and a total of 8 sessions will be conducted at the chosen intervention centre from April 2019 to May 2019. The main study will be one year from April 2019 to April 2020. The intervention will occur in both individual and group settings. 2 to 4 students will be allocated to each individual session, and others will attend the group sessions. The project team will be made up of many professional including a qualified AAI dog, qualified AAI dog handler, occupational therapist, pediatrician, clinical psychologist, speech therapist, school teacher or school social worker. The pediatrician, clinical psychologist and speech therapist will conduct a pre- and post-evaluation by assessing the child's condition before and after the programme. The speech therapist will supervise the therapy session in place of the occupational therapist if there is a speech impediment in the participant. The activities carried out during the intervention were previously planned by the project team members, who chose among the following per appropriateness for each session and depending on the interests of the subject: 1) sensorial and upper limb stimulation (brush, pet, and play fetch with the dog); 2) training on activities of daily living (give water and food to the dog) and gait (walking with the dog); 3) socialization and recreation (dog show; playing with the dog's supplies; dog drawing; agility courses-guide the dog through obstacles such as cones and ropes; dog clothes-form words that express feelings and attach them to the dog clothes with Velcro; stories about the dog-daily routine, origin). Before the start of the first session, the participants and their caregivers will complete the instruments described below with the help of a member of the research team trained for this purpose. At the end of the programme, the participants and their caregivers will fill out the same instruments again, and the physiological parameters will be re-measured. Outcome measuresments include problem identification, effectiveness of AAI, changes in quality of life, benefits and limitations of this intervention, and cost and feasibility of implementing the Animal Assisted Intervention Dog Traing Programme in Hong Kong which includes the cost of transport, and the cost of AAI dog and dog handler training.

ELIGIBILITY:
Inclusion Criteria:

-Either gender aged 6 to 18 years old; have mild to moderate autism

Exclusion Criteria:

-Who are not interested in the intervention and/or afraid of animals; who are allergic to animals; with severe mental/cognitive issues that might lead to injuries/ inconvenience to the animals and increase the likelihood of undersired events

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | within two weeks Pre-treatment and within two weeks Post-treatment
  The Strengths and Difficulties Questionnaire (SDQ) is a common tool used to screen behavior in children and teenagers aged 3-16 years. It looks at emotional and behavioral challenges in five areas: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Parents, teachers, or the young person themselves usually complete the 25-question survey. The responses help identify strengths and difficulties in different aspects. The SDQ is employed in clinics, research, and schools to spot children at risk of emotional or behavioral issues and track progress in intervention programs. Based on the scoring of SDQ, 80% of children scored normal, 10% borderline, and 10% abnormal.
Pediatric Quality of Life Inventory (PedsQL) 4.0 Core | within two weeks Pre-treatment and within two weeks Post-treatment
  The Pediatric Quality of Life Inventory (PedsQL) 4.0 Core is a questionnaire used to assess the well-being of children and teenagers. It looks at their physical, emotional, social, and school functioning. Kids aged 2-18 years can fill it out, as well as their parents or caregivers. The results give a detailed picture of the child's quality of life. This tool is valuable in clinics, research, and schools to understand how health issues or treatments affect a child's overall happiness and health. The PedsQLTM 4.0 Generic Core Scales use a scale from 0-100, where higher scores mean better Health-Related Quality of Life. To calculate scores, reverse score the items on a 0-4 scale to a 0-100 scale: 0=100, 1=75, 2=50, 3=25, 4=0.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Wilfred Wong, p.hD. In Public Health, Principal Investigator — Department of Paediatrics & Adolescent Medicine, The University of Hong Kong
Locations (1):
- Special Schools in Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] First MB. Diagnostic and statistical manual of mental disorders, 5th edition, and clinical utility. J Nerv Ment Dis. 2013 Sep;201(9):727-9. doi: 10.1097/NMD.0b013e3182a2168a. No abstract available. PMID 23995026
- [Background] Winkle M, Crowe TK, Hendrix I. Service dogs and people with physical disabilities partnerships: a systematic review. Occup Ther Int. 2012 Mar;19(1):54-66. doi: 10.1002/oti.323. Epub 2011 Aug 19. PMID 21858889
- [Background] Hall SS, Wright HF, Mills DS. What Factors Are Associated with Positive Effects of Dog Ownership in Families with Children with Autism Spectrum Disorder? The Development of the Lincoln Autism Pet Dog Impact Scale. PLoS One. 2016 Feb 19;11(2):e0149736. doi: 10.1371/journal.pone.0149736. eCollection 2016. PMID 26894820
- [Derived] Wong WHS, Chen C, Tso A, So HK, Wong JPY, Tinsley H, Chung CHY, Luk RKW, Ip P. Dog-assisted therapy on Hong Kong children with autism spectrum disorder: an exploratory randomized controlled trial. Eur J Pediatr. 2026 Jan 9;185(1):64. doi: 10.1007/s00431-025-06720-6. PMID 41511681